CLINICAL TRIAL: NCT05132881
Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation (TAVNS) on Anxiety and Brain Function in Distressed Healthcare Professionals
Brief Title: Effect of (TaVNS) on Anxiety and Brain Function in Distressed Health Care Workers
Acronym: fMRIVNS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Andrew Newberg, Professor, Department of Integrative Medicine and Nutritional Sciences; Professor, Department of Radiology, Thomas Jefferson University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 221D.069
Record Dates: First submitted 2021-10-21; First posted 2021-11-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Distress, Emotional; Effects of Vibration; Healthy
Keywords: Vagal Nerve Stimulation; Distressed Workers; Work-related Stress; Magnetic Resonance Imaging (MRI); Functional Magnetic Resonance Imaging (fMRI); Healthy Controls
MeSH Terms: conditions — Anxiety Disorders; Occupational Stress

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned by randomization to place individuals into the TaVNS or wait-list groups using a permuted block design with a 1:1 ratio to the group assignments. Subjects will be assigned a study number that will be used on the research files. Each subject will be informed of their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Transcutaneous Auricular Vagal Nerve Stimulation Intervention Group Distressed Healthcare Workers (Active Comparator): Two subgroups will be included in fMRI in the Active Comparator Group where scans performed during the initial evaluation period (pre) and at 3 months (post). Subgroup I of 30 subjects will undergo fMRI scans that will include structural imaging and functional imaging with Blood Oxygen Level Dependent Imaging (BOLD) scan and two arterial spin labeling (ASL) scans. This same imaging protocol, which takes a total of about 45 minutes, will be performed initially and then after the 3 month TaVNS program or the waitlist period. All scans will be co-registered and comparable slices of the cerebral cortex will be examined.
  Subgroup II will consist of 10 study subjects all receiving the TaVNS program who will undergo fMRI initially and then again at 3 months. This group will be scanned while wearing the TaVNS system (a special one that can be used in the MRI environment) and the fMRI will be used to evaluate the direct effects of the TaVNS while turned on and off in the scanner.
  Interventions: Other: Neuvana 2.0 Transcutaneous Auricular Vagal Nerve Stimulation (TaVNS)
- Waitlist Control Distressed Healthcare Workers Delayed TaVNS Group (Active Comparator): After baseline and 3 month imaging is completed. The waitlist control subgroups will be included in fMRI scans performed during the initial evaluation period (pre) and at 3 months (post). Subgroup I of 30 subjects will undergo fMRI scans that will include structural imaging and functional imaging with Blood Oxygen Level Dependent (BOLD) scan and two arterial spin labeling (ASL) scans. a typical morning waking up). This same imaging protocol, will be performed initially and then after the 3 month waitlist period. All scans will be co-registered and comparable slices of the cerebral cortex will be examined. After the waitlist imaging is completed the subjects will be offered the TaVNS health device.
  Interventions: Other: Waitlist Control
- Healthy Controls: Group II and III (Other): The Investigators will also plan to recruit 10 healthy controls with no reports of psychological distress (i.e. less than 2 on the SUDS). These 10 healthy controls will have the TaVNS placed while receiving two fMRI scans approximately 3 months apart. These control subjects will be used to compare the subgroup of study subjects to ensure that any changes are not associated with test-retest effects.the Investigators also plan to recruit 50 additional healthy controls with no reports of psychological distress (i.e. less than 2 on the SUDS.) These 50 controls will have the TaVNS placed while receiving one fMRI scan sequence in one day while wearing a non-metalllic set of the TaVNS ear buds to evaluate the effects of the functional changes that may occur in the brain while using the TaVNS device.
  Interventions: Other: Healthy Controls: Substudy Group III; Other: Distressed Workers: Subgroup II

INTERVENTIONS:
Other: Neuvana 2.0 Transcutaneous Auricular Vagal Nerve Stimulation (TaVNS) — The intervention administered is the TaVNS program and the fMRI scans to evaluate changes in the brain. The TaVNS program consists of placing ear buds from the device into each ear. They are initially sprayed once with a small amount of saline that is also provided as part of the TaVNS materials. Once the ear buds are placed in each ear, the test subject will start a preprogramed session of vibrations that will stimulate the vagus nerve. The session will last for 15 minutes and then the subject will take the ear buds out and clean them. They will use the TaVNS program once a day for 3 months.
  Other Names: Active TaVNS Program in Distressed Workers
  Arms: Transcutaneous Auricular Vagal Nerve Stimulation Intervention Group Distressed Healthcare Workers
Other: Waitlist Control — Baseline imaging and follow up imaging for comparison to the TaVNS health device group at approximately 3 months. The TaVNS intervention is offered after completion of the imaging.
  Other Names: Waitlist Control Group of Distressed Workers
  Arms: Waitlist Control Distressed Healthcare Workers Delayed TaVNS Group
Other: Healthy Controls: Substudy Group III — fMRI Imaging to evaluate the effects of the functional changes that may occur in the brain while using the TaVNS device during one fMRI session.
  Other Names: Controls without Distress for one fMRI imaging session while using the TaVNS health device
  Arms: Healthy Controls: Group II and III
Other: Distressed Workers: Subgroup II — Subgroup II of 10 subjects with distress(all receiving TaVNS) will undergo fMRI scans with the TaVNS system being turned on and off while in the scanner to observe for any immediate effects and to evaluate the effects of the functional changes that may occur in the brain while using the TaVNS device during one fMRI session.
  Other Names: Distressed Workers for fMRI one fMRI imaging while using the TaVNS health device
  Arms: Healthy Controls: Group II and III

SUMMARY:
The purpose of this research is to measure alterations in anxiety and brain activity associated with the use of an approved health device called Transauricular Vagal Nerve Stimulation (TaVNS) in distressed persons who work in a health care and distressed healthcare workers in the the Philadelphia, PA region. The Investigators will be using functional magnetic resonance imaging (or fMRI) to measure changes in each subject's brain function during the use of VNS. This study is designed to allow researchers to understand the changes in cerebral (brain) activity that occur when a subject uses VNS. Thus, the primary goal of the proposed study is to evaluate the ability of the TaVNS system to reduce distress and change neurophysiology among health care providers.

The Investigators, hypothesize that using the TaVNS device will help reduce distress in individuals.

In order to understand the mechanisms of change that occur while using the VNS study, the Investigators have added a substudy of participants who do not experience high levels of distress to evaluate the effects of the functional changes that may occur in the brain while using the TaVNS device.

In addition to the primary aims of the overalll study to assess distress in workers while enrolled in a TaVNS program, a subgroup of 50 subjects will undergo functional magnetic resonance imaging (fMRI) while using the VNS device to assess the changes in the brain including neurophysiological effects of TaVNS.

The goal of this substudy is to observe the changes in the brain while using the TaVNS earbuds in the MRI to increase our understanding of the mechanisms and processing involved while using TaVNS. In this substudy, which is amendment version 3.0, the investigators have increased the number of persons to include 50 subjects who will use the device in the MRI to evaluate the neural processes and cerebral blood flow while using TaVNS.

DETAILED DESCRIPTION:
A total of up to 90 distressed persons who work in health care and health care providers in the Philadelphia, PA region, will be screened for this study. From that group, the researchers plan to enroll enough subjects to have 80 fully complete the study. The 90 screened subjects will allow for screen failures and subjects who withdraw early from the study. All subjects will receive an initial evaluation using symptom questionnaires (these will include the Global Severity Index of the Brief Symptom Inventory-18 which is the primary outcome, and secondary outcomes as measured by the Maslach Burnout Scale, GAD-7 (anxiety), PHQ-9 (depression), the Connor Davidson Resilience Scale-25 (CD-RISC), and the Insomnia Severity Index (ISI) and physiological measures that will consist of heart rate variability (HRV) and galvanic skin resistance (GSR). Subjects will then be randomized to either the 3 month TaVNS program or the 3 month waitlist group. At one month, subjects will receive a follow up request to complete the same questionnaires as in the initial evaluation for an interim evaluation. Then after receiving the TaVNS program or being in the waitlist control group for 3 months, the subjects will have a repeat of the questionnaires and physiological testing. Subjects in the waitlist group will then be provided the TaVNS program to be used for 3 months. This group will be asked to complete one final set of symptom questionnaires at the completion of using the TaVNS program.

Two subgroups will be included in fMRI scans performed during the initial evaluation period (pre) and at 3 months (post). Subgroup I of 30 subjects (15 in TaVNS group and 15 in waitlist control) will undergo fMRI scans that will include structural imaging and functional imaging with Blood Oxygen Level Dependent Imaging (BOLD) scan and arterial spin labeling (ASL) scans. Specifically, during the ASL scans (each approximately 5 minutes long), a script of the subject's most distressing recollection(s) will be read from an audio file script while each subject is in the MRI scanner. Changes in brain function will be compared between the stress script and a neutral script (that describes a typical morning waking up). This same imaging protocol, which takes a total of about 45 minutes, will be performed initially and then after the 3 month TaVNS program or the waitlist period. All scans will be co-registered and comparable slices of the cerebral cortex will be examined.

Subgroup II will consist of 10 study subjects all receiving the TaVNS program who will undergo fMRI initially and then again at 3 months. This group will be scanned while wearing the TaVNS system (a special one that can be used in the MRI environment) and the fMRI will be used to evaluate the direct effects of the TaVNS while turned on and off in the scanner. The imaging protocol will take a total of about 45 minutes. In addition to the 10 study subjects, the researchers will also plan to recruit 10 healthy controls with no reports of psychological distress (i.e. less than 2 on the SUDS). These 10 healthy controls will have the TaVNS placed while receiving two fMRI scans approximately 3 months apart. These control subjects will be used to compare the subgroup of study subjects to ensure that any changes are not associated with test-retest effects.

The subgroups will be filled with eligible and interested subjects. If the subject is interested and is able to undergo fMRI scanning, the subject will be placed in Subgroup I until enrollment is filled and then subsequently subjects will be enrolled into Subgroup II until enrollment is filled. Any eligible subject that is unwilling or unable to undergo fMRI scanning will be placed in the general, non-scanning group. Once the two subgroups are filled, any remaining eligible subjects will be placed in the general, non-scanning group.

Substudy:

A total of 50 additional subjects will be screened to receive one MRI imaging while using the TaVNS earbuds. Subjects who are eligible to receive an MRI scan will be enrolled from the geographical region. Participants may also be self-referred by responding to flyers to inquire more about the study. The objective of the substudy (Subgroup III) is to increase our understanding of the mechanisms and neurophysiological response while using the TaVNS in the MRI scanner by evaluating cerebral blood and activation states while the TaVNS is "on" and "off" during a single fMRI session while using the TaVNS.

Endpoints for the Imaging Using TaVNS Substudy

A substudy (Subgroup III) of 50 subjects, with no randomization, will undergo fMRI scans with the TaVNS system being turned on and off while in the scanner to observe for any immediate effects. While the system is generally not supposed to be used in the MRI environment, a special non-magnetic version (that can be used in the MRI environment) will be used to test this change. Specifically, the unit itself will be outside of the MRI environment and will be attached to the earbuds using a non-magnetic wire.

Secondary Endpoints:

Secondary endpoints may include clinical measures including the Maslach Burnout Scale, GAD-7 (anxiety), PHQ-9 (depression), Connor Davidson Resilience Scale-25 (CD-RISC), Insomnia Severity Index (ISI), and physiological measures that will consist of heart rate variability (HRV) and blood pressure.

Additional secondary endpoints will be the baseline fMRI scans that will include structural imaging and functional imaging with Blood Oxygen Level Dependent Imaging (BOLD) scan and two arterial spin labeling (ASL) scans. fMRI scan data for this substudy may be compared between the MRI Imaging group and the TaVNS group and waitlist control.

Subgroup II will consist of 10 study subjects all receiving the TaVNS program who will undergo fMRI initially and then again at 1 month (+30 days). This group will be scanned while wearing the TaVNS system (a special one that can be used in the MRI environment) and the fMRI will be used to evaluate the direct effects of the TaVNS while turned on and off in the scanner. The imaging protocol will take a total of about 45 minutes.

In addition to the 10 study subjects in the distressed workers group, we intend to recruit 50 healthy controls with no reports of psychological distress (i.e. less than 2 on the SUDS) with no biofeedback evaluation. These 50 healthy controls will have the TaVNS placed while receiving one fMRI scans. These control subjects will be used to compare the subgroup of study subjects to understand the changes in the brain while using the TaVNS. These participants will be consented with an informed consent form that describes the substudy in more detail. Subjects in the substudy Group III will receive only one fMRI imaging session on one day and will be asked to complete surveys. Participants in this substudy will have heart rate collected at baseline, during and after the fMRI while using the VNS.

All subjects will receive an initial evaluation using symptom questionnaires (these will include the Global Severity Index of the Brief Symptom Inventory-18 which is the primary outcome, and secondary outcomes as measured by the Maslach Burnout Scale, GAD-7 (anxiety), PHQ-9 (depression), the Connor Davidson Resilience Scale-25 (CD-RISC), and the Insomnia Severity Index (ISI).

The eligibility for imaging is the same for all groups with the exception of Subjective Units of Distress Scores.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female persons who work in health care and health care workers (all races and ethnicity) >21 years of age
2. All subjects must have a smartphone device that can be used in conjunction the Neuvana 2.0
3. Drug-free from medications that may affect brain physiology such that the imaging results will not be useful as determined by the PI.
4. Able to understand and provide signed informed consent. Available and willing to be followed -up according to study protocol
5. Female subjects of childbearing potential have a negative pregnancy test
6. Subjects have no significant medical neurological or psychological disorders
7. Stable health problems that should have no substantial effect on cerebral blood flow will be allowed (i.e. controlled hypertension, medication controlled diabetes).
8. Current medications and supplements will be reviewed by the Principal Investigator or a designated physician or health practitioner. Subjects may take medications or supplements but should be on a stable dose regimen for at least 3 months. For those receiving TaVNS program, it is preferable that subjects remain on that dose for the full TaVNS program period (with the exception of having an adverse reaction in which the medication or supplement must be stopped).
9. PI will evaluate each subject for any potential medical issues that might be a problem and will consult with the subject's primary care provider if there are any questions about it.

Additional Inclusion Criteria for the TaVNS program for Distressed Workers

1. Distress scored as at least a 6 or greater on the SUDS distress level from 1 to 10.
2. Distressing recollection(s) that causes physiological reactivity (i.e., increased heart rate and/or increased skin conductance level - SCL), as described above.

Healthy control with no distress or other exclusion criteria

Exclusion Criteria:

1. Any medical conditions that may interfere with cerebral blood flow as determined by the PI.
2. Currently taking medication that might affect cerebral blood flow as per the P.I. (i.e. antidepressants, antipsychotics, anxiolytics, benzodiazepines, sedatives, anti-seizure medications, but with the exception of those described above)
3. Subject is unable or unwilling to lie still in the scanner (i.e. due to claustrophobia or weight)
4. Subject has metal in their body or other reason that they cannot undergo magnetic resonance imaging.
5. Previous brain surgery or intracranial abnormalities they may complicate interpretation of the brain scans (e.g., stroke, tumor, vascular abnormality).
6. Pregnancy or breastfeeding
7. Concurrent participation in another research protocol that might affect the outcome of this study.
8. Use of a defibrillator or pacemaker or other implanted or metallic electronic device. Doing so could cause electric shock, burns, electrical interference, or death.
9. Epilepsy
10. History of Seizures
11. Temporomandibular Joint Disorder, Bell's Palsy, impaired cranial nerve function, or facial pain.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Subjective Units of Distress Survey | Screening Measure Subjects will be evaluated at baseline.
  The Subjective Units of Distress Survey (SUDS) is a way for participants to communicate how much distress they are currently feeling using a 0 to 10 scale with zero corresponding to a relaxed state without distress and ten corresponding to extreme distress filled with panic, tension, fear, and anxiety.
Subjective Units of Distress Survey | Change from baseline and after using the TaVNS system approximately 90 days (~3 months)] .
  The Subjective Units of Distress Survey (SUDS) is a way for participants to communicate how much distress they are currently feeling using a 0 to 10 scale with zero corresponding to a relaxed state without distress and ten corresponding to extreme distress filled with panic, tension, fear, and anxiety.
Subjective Units of Distress Survey | Evaluate at baseline to evaluate distress for healthy controls in Group III
  The Subjective Units of Distress Survey (SUDS) is a way for participants to communicate how much distress they are currently feeling using a 0 to 10 scale with zero corresponding to a relaxed state without distress and ten corresponding to extreme distress filled with panic, tension, fear, and anxiety.
Heart Rate Variability for Active and Waitlist | Screening Measure Subjects will be evaluated at baseline
  Heart rate variability (HRV) is the physiological phenomenon of the variation in the time interval between consecutive heartbeats in milliseconds.
Heart Rate Variability for Active and Waitlist | Change from baseline and after using the TaVNS system approximately 90 days (~3 months)] .
  Heart rate variability (HRV) is the physiological phenomenon of the variation in the time interval between consecutive heartbeats in milliseconds.
Galvanic Skin Resistance (GSR) for Active and Waitlist | Screening Measure Subjects will be evaluated at baseline
  To measure changes in sweat gland activity, which reflect the intensity of participants' emotional state
Galvanic Skin Resistance (GSR) for Active and Waitlist | Change from baseline and after using the TaVNS System approximately 90 days (~3 months)]
  To measure changes in sweat gland activity, which reflect the intensity of participants' emotional state
Functional magnetic resonance imaging (fMRI) in all groups | Subjects will be evaluated at baseline
  This scan will be used to assess functional connectivity, tractography, and brain volume
Functional magnetic resonance imaging (fMRI) in Active and Waitlist Groups | Change from baseline and after using the TaVNS system approximately 90 days (~3 months)] .
  This scan will be used to assess functional connectivity, tractography, and brain volume
Blood Oxygen Level Dependent Imaging scan in all groups | Subject will be evaluated at baseline
  Blood Oxygen Level Dependent Imaging (BOLD) scan analysis, used to observe different areas of the brain or other organs, which are found to be active at any given time.
Blood Oxygen Level Dependent Imaging scan in Active and Waitlist Groups | Change from baseline and after using the TaVNS System approximately 90 days (~3 months)]
  Blood Oxygen Level Dependent Imaging (BOLD) scan fMRI analysis, used to observe different areas of the brain or other organs, which are found to be active at any given time.
Arterial spin labeling scan in all groups | Subjects will be evaluated at baseline
  Arterial spin labeling (ASL) scan fMRI analysis, used to quantify cerebral blood perfusion by labelling blood water as it flows throughout the brain.
Arterial spin labeling scan in Active and Waitlist Groups | Change from baseline and after using the TaVNS System approximately 90 days (~3 months)]
  Arterial spin labeling (ASL) scan fMRI analysis used to quantify cerebral blood perfusion by labelling blood water as it flows throughout the brain.

SECONDARY OUTCOMES:
The Maslach Burnout Scale | Subjects will be evaluated at baseline with questionnaires.
  To measure feelings of being emotionally overextended and exhausted for health care professionals.The higher the score in each subgroup, the higher the emotional exhaustion and depersonalization, or the lower the sense of personal accomplishment.
The Maslach Burnout Scale | Subjects will be evaluated at approximately three months follow up with questionnaires.
  To measure feelings of being emotionally overextended and exhausted for health care professionals.The higher the score in each subgroup, the higher the emotional exhaustion and depersonalization, or the lower the sense of personal accomplishment.
The Maslach Burnout Scale | Subjects will be evaluated approximately six months follow up with questionnaires.
  To measure feelings of being emotionally overextended and exhausted for health care professionals. The higher the score in each subgroup, the higher the emotional exhaustion and depersonalization, or the lower the sense of personal accomplishment.
Patient Health Questionnaire | Subjects will be evaluated at baseline with questionnaires.
  Patient Health Questionnaire (PHQ-9)(depression) is the depression module to monitor the severity of depression and response to treatment. The range of the possible scores for the PHQ-9 are 0-27 with higher scores for worse symptoms.
Patient Health Questionnaire | Subjects will be evaluated at approximately three months follow up with questionnaires.
  Patient Health Questionnaire (PHQ-9)(depression) is the depression module to monitor the severity of depression and response to treatment. The range of the possible scores for the PHQ-9 are 0-27 wither higher scores for worse symptoms.
Patient Health Questionnaire (PHQ-9)(depression) | Subjects will be evaluated at baseline and approximately six months follow up with questionnaires.
  Patient Health Questionnaire (PHQ-9)(depression) is the depression module to monitor the severity of depression and response to treatment.The range of the possible scores for the PHQ-9 are 0-27 with higher scores for worse symptoms.
General Anxiety Disorder | Subjects will be evaluated at baseline with questionnaires.
  The General Anxiety Disorder (GAD-7) is a valid tool for screening for General Anxiety Disorder and assessing its severity. The GAD-7 consists of 7 questions that correspond to scores of anxiety. The range of scores is from 0 to 21; a higher score indicates greater anxiety.
General Anxiety Disorder | Subjects will be evaluated at baseline and approximately three months follow up with questionnaires.
  The General Anxiety Disorder (GAD-7) is a valid tool for screening for General Anxiety Disorder and assessing its severity. The GAD-7 consists of 7 questions that correspond to scores of anxiety. The range of scores is from 0 to 21; a higher score indicates greater anxiety.
General Anxiety Disorder | Subjects will be evaluated at baseline and approximately six months follow up with questionnaires.
  The General Anxiety Disorder (GAD-7) is a valid tool for screening for General Anxiety Disorder and assessing its severity. The GAD-7 consists of 7 questions that correspond to scores of anxiety. The range of scores is from 0 to 21; a higher score indicates greater anxiety.
Connor Davidson Resilience Scale-25 (CD-RISC) | Subjects will be evaluated at baseline with questionnaires.
  The Conner Davidson Resilience Scale-25 (CD-RISC-25) consists of 25 questions. The range of possible scores is 0-100 with a higher score indicating a higher chance of resiliency. The Connor-Davidson Resilience Scale is a test that measures resilience or how well one is equipped to bounce back after stressful events, tragedy, or trauma.
Connor Davidson Resilience Scale-25 | Subjects will be evaluated at approximately three months follow up with questionnaires.
  The Conner Davidson Resilience Scale-25 (CD-RISC-25) consists of 25 questions. The range of possible scores is 0-100 with a higher score indicating a higher chance of resiliency. The Connor-Davidson Resilience Scale is a test that measures resilience or how well one is equipped to bounce back after stressful events, tragedy, or trauma.
Connor Davidson Resilience Scale-25 | Subjects will be evaluated at baseline and approximately six months follow up with questionnaires.
  The Conner Davidson Resilience Scale-25 (CD-RISC-25) consists of 25 questions. The range of possible scores is 0-100 with a higher score indicating a higher chance of resiliency. The Connor-Davidson Resilience Scale is a test that measures resilience or how well one is equipped to bounce back after stressful events, tragedy, or trauma.
Insomnia Severity Index | Subjects will be evaluated at baseline with questionnaires.
  The Insomnia Severity Index (ISI) is a brief instrument comprised of 7 questions designed to assess the severity of both nighttime and daytime components of insomnia. The scores are rated 0-28 with higher scores corresponding to more sleep difficulties.
Insomnia Severity Index | Subjects will be evaluated at baseline and approximately three months follow up with questionnaires.
  The Insomnia Severity Index (ISI) is a brief instrument comprised of 7 questions designed to assess the severity of both nighttime and daytime components of insomnia. The scores are rated 0-28 with higher scores corresponding to more sleep difficulties.
Insomnia Severity Index | Subjects will be evaluated at baseline and approximately six months follow up with questionnaires.
  The Insomnia Severity Index (ISI) is a brief instrument comprised of 7 questions designed to assess the severity of both nighttime and daytime components of insomnia. The scores are rated 0-28 with higher scores corresponding to more sleep difficulties.
Global Severity Index of the Brief Symptom Inventory-18 | Subjects will be evaluated at baseline .
  The Brief Symptom Inventory (BSI-18) is a brief self-report survey to assess the extent of distress or annoyance. Responses were rated ranging from 1 to 5 for a total score of 18-90. A higher score indicates greater distress or annoyance.
Global Severity Index of the Brief Symptom Inventory-18 | Subjects will be evaluated at three months after using the TaVNS system.
  The Brief Symptom Inventory (BSI-18) is a brief self-report survey to assess the extent of distress or annoyance. Responses were rated ranging from 1 to 5 for a total score of 18-90. A higher score indicates greater distress or annoyance.
Global Severity Index of the Brief Symptom Inventory-18 | Subjects will be evaluated at six months after using the TaVNS system.
  The Brief Symptom Inventory (BSI-18) is a brief self-report survey to assess the extent of distress or annoyance. Responses were rated ranging from 1 to 5 for a total score of 18-90. A higher score indicates greater distress or annoyance.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Newberg, Principal Investigator — Department of Integrative Medicine and Nutritional Sciences
Locations (1):
- Thomas Jefferson University, Marcus Institute of Integrative Health Centers, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
After each participant completes the study, study scan data will be shared with co-investigators; participants may receive a copy of each scan after study completion.
Supporting Information: CSR
Time Frame: Study scan report will be offered to the subject after subject completes study
Access Criteria: Access only to authorized research staff and study participants